CLINICAL TRIAL: NCT05226559
Title: Effectiveness of Multimodal Physical Therapy for Episodic and Chronic Migraine With Concomitant Cervical Musculoskeletal Dysfuntions: Randomized Clinical Trial
Brief Title: Effectiveness of Multimodal Physical Therapy in Migraine
Acronym: MIGPHYSTREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Armando Perrotta, Principal Investigator, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIGRA012021
Record Dates: First submitted 2022-01-11; First posted 2022-02-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Migraine; Musculoskeletal Neck Pain; Musculoskeletal Disorder of the Neck; Chronic Migraine; Episodic Migraine
Keywords: Migraine;; Chronic Migraine;; Physical Therapy;; Cervical musculoskeletal dysfunction;; Joint Dysfunction;; trigger point
MeSH Terms: conditions — Migraine Disorders; Joint Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, parallel group, randomized clinical trial.
Who Masked: Care Provider, Investigator
Masking Description: Physiotherapists are blinded toward the diagnosis and outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Physical therapy approach plus usual care (Active Comparator): HVLA spinal manipulation, mobilization, soft tissue treatment, therapeutic exercise, education, plus standard pharmacological treatment.
  Interventions: Procedure: Multimodal Physical therapy approach plus usual care; Drug: Usual care
- Usual care (No Intervention): Standard pharmacological treatment alone

INTERVENTIONS:
Procedure: Multimodal Physical therapy approach plus usual care — HVLA spinal manipulation, mobilization, soft tissue treatment, therapeutic exercise, education, plus standard pharmacological treatment.
  Other Names: Intervention group
  Arms: Multimodal Physical therapy approach plus usual care
Drug: Usual care — Standard pharmacological treatment alone.
  Other Names: Usual care group
  Arms: Multimodal Physical therapy approach plus usual care

SUMMARY:
INTRODUCTION: It is very common that migraine patients could refer neck pain during or after the pain phase of migraine, suggesting that migraine pathophysiological mechanisms could be effective in activating neck pain pathways and be part of the migraine attack. Due to the therapeutic effect of multimodal physical therapy (mobilization and/or manipulation plus exercises) on several pain conditions arising from articular and/or muscular structures such as neck pain, and given the close clinical, anatomical and pathogenetic bi-directional relationship between neck pain and migraine, it would be of interest to evaluate the effectiveness of the physical treatment of the neck region in migraine pain.

PURPOSE: to evaluate the efficacy of a combined multimodal physical therapy approach plus usual care vs. usual care alone in subjects with episodic and chronic migraine with concomitant cervical musculoskeletal dysfunctions.

STUDY DESIGN: this is a prospective, parallel group, randomized clinical trial. METHODS: A total of 56 subjects aged 18-65 who meet criteria for episodic or chronic migraine with concomitant cervical musculoskeletal dysfunctions will be randomly assigned to receive, musculoskeletal focused multimodal physical therapy (16 sessions over 8 weeks) plus usual care treatment vs. usual care alone.

CONFLICT OF INTEREST: not declared.

DETAILED DESCRIPTION:
Study design This is a prospective, parallel group, randomized clinical trial evaluating multimodal care plus usual care vs. usual care alone in episodic and chronic migraine with concomitant muscoloskeletal dysfunctions.

The total study duration from the Screening Visit to the Completion Visit is approximately 28 weeks and includes a Screening Period (12 weeks) and an intervention period (8 weeks) followed by an observational period post treatment (8 weeks) for each participant.

Procedures Eligible patients who provided informed consent started the screening period of 12 weeks to confirm migraine frequency, stable prophylactic migraine treatment, including and inclusion/exclusion criteria. During the screening period patients collected informations including number of monthly migraine days, use of acute medication, migraine days with use of acute medication, headache severity (graded as mild, moderate or severe) and duration by using daily migraine report. Migraine associate disability (MIDAS), neck associated disability (NDI) and level of depression (PHQ-9) were detected by using appropriate tests at the end of the 12-week screening period (week 12), at the end of the 8-week intervention period (week 20), and at the end of the study 8 weeks after the last treatment (week 28). During the screening period each participant underwent a physical examination test by physical therapists (LDA, FL, MS) specialized in manual therapy to detect cervical musculoskeletal dysfunctions, including temporomandibular disorders, which are potentially tractable with physical therapy. Physical examination assessed cervicothoracic spine posture, ranges of motion, presence of myofascial trigger points, cervical and temporo-mandibular joint movement restriction.

Procedures Participants who have completed the screening period will be randomized 1:1, using an automatic allocation system, to receive multimodal physical therapy treatment in addition to standard pharmacological treatment or standard pharmacological treatment alone (usual care). The sample will be stratified according to the diagnosis of headache (episodic migraine or chronic migraine), cervical and / or temporomandibular musculoskeletal dysfunction and concomitant myofascial disorder. After 8 weeks of treatment, participants will be monitored for a follow-up phase free of physical treatment lasting an additional 8 weeks.

A research assistant in the study (NM) will monitor the blinding of the study and assign the participants to the intervention.

The physical therapist and the neurologist will be blinded each other in relation to the diagnosis of headache and the type physical therapy treatment that will be practiced on the patient.

Examination procedures

Functional evaluation of the cervical spine

* Cervical active (CROM) and passive (PROM) movements (flexion, extension, rotation, anteposition and retroposition of the head), the results will be recorded with presence / absence (YES 1 / NO 0) of hypomobility and / or evocation of pain. The overall result will be the combined hypomobility and pain scores for both sides;
* Flexion Rotation Test (FRT) for the presence of pain, hypomobility and degrees of movement (> 32).
* Palpation of trigger points (TP): trigger points are defined as a painful point on palpation at a muscle belly, recognized by the patient as the usual headache (active trigger point) or referred to a region not related to the usual headache localization (latent trigger point). Four TPs will be explored in the sternal portion of the sternocleidomastoid muscle, 4 TP in the masseter muscle, 3 TP in the temporal muscle, 2 TP in the suboccipital muscles, 4 TP in the trapezius muscle. The number of active and latent trigger points will be recorded. The total score will be the combined number of active and latent trigger points for both sides.
* Passive accessory intervertebral movements (PAIVMs): central and unilateral antero-posterior movement at C0-3. The number of low-mobility and / or painful joints and directions of movement will be recorded. The total score will be the number of low-mobility and painful joints combined. Reproduction and resolution: unilateral postero-anterior movement supported at C0-3. If there will be reproduction and resolution of headache symptoms, it will be assigned a value of 1.
* Chest screening (T1-T6): active right and left rotation with arms crossed over the chest (standardized) and head looking forward; manual palpation of the posterior-anterior, central and unilateral joint . Results will be recorded with presence / absence (YES 1 / NO 0) of hypomobility and / or evocation of pain. The overall result will be the combined hypomobility and pain score for both sides. The number of clinical signs will be recorded (maximum 5 per vertebral segment: right / left rotation, central PA, unilateral right / left PA).
* Cervical rotation lateral flexion test C7-T1-K1 (CRLFT): evaluates the mobility or the presence of an elevated position of the first rib (K1) in the combined contralateral rotation movement combined with ipsilateral lateral flexion to the side of the rib to be evaluated .
* Cranio Cervical Flexion Test (CCFT): is a test for the evaluation of the deep cervical flexor muscles using the STABILIZER Biofeedback. The pressure biofeedback value varies between 20 and 28 mmHg; The test consists in maintaining the contraction for 10 seconds without compensation of the superficial muscles. The mmHg value will be recorded and held for 10 seconds without compensation.
* Temporomandibular joint evaluation
* Evaluation of temporomandibular joint noise: it is performed using a stethoscope and evaluating the right and left joint noises.
* The temporomandibular joint will be palpated bilaterally to assess the presence of tenderness, pain, swelling and assessment of movement patterns. Any anomaly will be noted as presence / absence (YES = 1, NO = 0).

Imaging and provocative maneuvers

* Cervical X-Ray
* MRI
* "Wainner Cluster"
* Evocation of the blink reflex

Interventions All visits and treatments will take place at the Headaches Medicine Unit of IRCSS Neuromed in Pozzilli (IS) and the study participants will be treated by three physical therapists: LD, MS, FL. All appointments by date and time will be recorded to monitor participants adherence to the treatment. The details of each individual treatment session, including any adverse effects related to the treatment, will be systematically recorded in the patient's medical record. Adverse events include: worsening of headache and / or neck pain and / or reduction of cervical joint ROM or any other health and safety event in relation to treatment.

The neurological and physical medicine examination, combined with the physical therapy evaluation, will include the complete history of the headache, evaluation of the risk factors that may indicate contraindication to the treatment, clinical history of the patient with particular focus on lifestyle habits and incorrect attitudes / postures that may promote musculoskeletal disorders and therefore pain, neck tension and headache.

Patients will receive a cycle of 16 sessions of multimodal physical therapy treatment in 8 weeks, followed by an 8-week suspension phase of the rehabilitation treatment. The first session and subsequent sessions including physical assessments (T1-T2) will have a duration of 50 minutes, all other sessions will have a duration of 30 minutes.

Multimodal physical therapy approach group

* Spinal manipulation therapy with HVLA (high velocity low amplitude) techniques that are able to reduce pain and improve the mobility of the manipulated joint with a consequent increase in the "range of motion". Furthermore, they have a series of neurophysiological effects of very high impact that occur locally and at a distance from the manipulated district. These techniques are able to raise the activation threshold of the stretch reflex of those myofascial tissues which, if they are in a spasm condition, can reduce the movement capacity of a joint district . The treated areas will be the upper cervical (C0-C3), the cervicothoracic junction (C7-T1-K1), the upper thoracic (T2-T4-K2) and the middle thoracic (T4-T6).
* The interventions also include spinal stabilization exercises shown during the treatment session, myofascial treatment techniques for soft tissues, joint mobilization and breathing and relaxation techniques, finally, changes in the ergonomics of the work and home environment will be recommended (tab2) and an illustrative brochure will be released containing management advice on migraine and the protocol of exercises to be performed at home. The average frequency of home exercises will be recorded during the sessions.

All these interventions will be shown and performed with the aim of improving the patient's self-efficacy in self-management of symptoms. The hypothesis is that manipulative manual therapy, combined with therapeutic exercise, may have a hypoalgesic effect in patients affects from migraine .

• Temporomandibular joint treatment: Treatment techniques consist of accessory (translational) movements of the temporomandibular region and / or techniques for the masticatory muscles, such as trigger point treatment and muscle stretching.

Statistical Analysis The calculation of the sample size was based on an effect size d = 0.5, 80% of the sample power and Bonferroni correction of the alpha to 0.05 for the main variable represented by the number of headache days per month. The total number of the sample was found to be 56 (28 subjects per group).

The differences between the data relating to the two groups of experimental and usual care treatment will be performed using ANOVA for repeated measures with Bonferroni correction p-value 0.05 for continuous variables and Kruskal-Wallis Test with correction by Dunn's Test for ordinal variables.

Risk of multimodal physical therapy approach

The risks of serious adverse events related to the multimodal physical therapy approach, including neurological and cerebrovascular diseases, are considered very low, however their exact incidence is unknown. Estimates range from 1 in 200,000 to 1 in several million cervical spine manipulations. Minor adverse events such as neck pain, stiffness, fatigue and headache are much more common in clinical practice. All participants were given instructions at the start of the study to report any adverse event (AE) to study staff within 24 hours. Safety measures included the occurrence of spontaneously reported treatment emergent adverse events.

ELIGIBILITY:
Inclusion criteria

* patients aged 18-65 years;
* patients with episodic migraine with and without aura (experiencing 6-14 days/month with migraine);
* patients with chronic migraine;
* patients who achieved >30% <50% reduction from their individual baseline in the number of monthly migraine days on therapy with standard stable pharmacological treatments during the past 3 months;
* concomitant cervical dysfunctions.

Exclusion criteria

* self-report of neck injury/trauma;
* acute radiculopathy;
* history of carotid or vertebral artery dissection;
* stroke;
* cervical/cranial nerve block in the past three months;
* pregnancy;
* history of infection;
* migraine attack during the assessment;
* diagnosis of other concomitant headaches (such as cervicogenic headache, tension-type headache, cluster headache, medication overuse headache);
* having received physical treatment in the past three months or botulinum toxin in the past six months;
* any unstable medical o psychiatric condition.
* history of any other rheumatic or chronic diseases such as fibromyalgia;
* neuralgias, or self-report of vestibular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in screening period monthly migraine days at the end of the intervention period (week 20) and at the end of the study (week 28) (daily migraine report) | At the end of the 12-week screening period (week 12), at the end of the 8-week intervention period (week 20), and at the end of the study 8 weeks after the last treatment (week 28)
  Number of monthly migraine days
Change in screening period monthly migraine days with use of acute medication at the end of the intervention period (week 20) and at the end of the study (week 28) (daily migraine report) | At the end of the 12-week screening period (week 12), at the end of the 8-week intervention period (week 20), and at the end of the study 8 weeks after the last treatment (week 28)
  Monthly migraine days with use of acute medication

SECONDARY OUTCOMES:
Change in screening period Migraine Disability Assessment Score (MIDAS) at the end of the intervention period (week 20) and at the end of the study (week 28) | At the end of the 12-week screening period (week 12), at the end of the 8-week intervention period (week 20), and at the end of the study 8 weeks after the last treatment (week 28)
  Migraine disability assessment score (MIDAS) The scale ranges between 0 "little or no disability" and 5 "severe disability"
Change in screening period Neck disability index (NDI) at the end of the intervention period (week 20) and at the end of the study (week 28) | At the end of the 12-week screening period (week 12), at the end of the 8-week intervention period (week 20), and at the end of the study 8 weeks after the last treatment (week 28)
  Neck disability index (NDI) Each of the 10 items is scored from 0 - 5. The score between 0 and 4 indicates "no disability", the score above 34 indicates a severe disability
Change in screening period Patient Health Questionnaire-9 (PHQ-9) at the end of the intervention period (week 20) and at the end of the study (week 28) | At the end of the 12-week screening period (week 12), at the end of the 8-week intervention period (week 20), and at the end of the study 8 weeks after the last treatment (week 28)
  Patient Health Questionnaire-9 (PHQ-9) The score between 0 and 4 indicates "none depression", the maximum score between 20 and 27 indicates a severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Armando Perrotta, MD, Principal Investigator — Neuromed IRCCS
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Ashina S, Bendtsen L, Lyngberg AC, Lipton RB, Hajiyeva N, Jensen R. Prevalence of neck pain in migraine and tension-type headache: a population study. Cephalalgia. 2015 Mar;35(3):211-9. doi: 10.1177/0333102414535110. Epub 2014 May 22. PMID 24853166
- [Background] Florencio LL, Chaves TC, Carvalho GF, Goncalves MC, Casimiro EC, Dach F, Bigal ME, Bevilaqua-Grossi D. Neck pain disability is related to the frequency of migraine attacks: a cross-sectional study. Headache. 2014 Jul-Aug;54(7):1203-10. doi: 10.1111/head.12393. Epub 2014 May 26. PMID 24863346
- [Background] Luedtke K, Starke W, May A. Musculoskeletal dysfunction in migraine patients. Cephalalgia. 2018 Apr;38(5):865-875. doi: 10.1177/0333102417716934. Epub 2017 Jun 22. PMID 28641450
- [Background] Bartsch T, Goadsby PJ. The trigeminocervical complex and migraine: current concepts and synthesis. Curr Pain Headache Rep. 2003 Oct;7(5):371-6. doi: 10.1007/s11916-003-0036-y. PMID 12946290